CLINICAL TRIAL: NCT01741584
Title: Effects of Physical Activity on the Brain in Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr. med. Agnes Floeel, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PA_memory_01
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stationary bike exercise (Experimental): 6 months of exercise (60% of anaerobic threshold)
  Interventions: Behavioral: stationary bike exercise
- aerobic (Placebo Comparator): 6 months of exercise <30% anaerobic threshold
  Interventions: Behavioral: aerobic

INTERVENTIONS:
Behavioral: stationary bike exercise
  Arms: stationary bike exercise
Behavioral: aerobic
  Arms: aerobic

SUMMARY:
The aim of the study is to investigate whether exercise improves cognitive and motor functions in Parkinson's disease. To test this hypothesis, the researchers study general brain functions in subjects with PD during a 6-months exercise program.

ELIGIBILITY:
Inclusion Criteria:

* UPDRS <15
* L-DOPA responsive
* <5 yrs since diagnosis

Exclusion Criteria:

* severe other diseases
* MMSE < 26
* treatment with psychiatric medication

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
UPDRS motor score | Prior to intervention and after 6 months of intervention

SECONDARY OUTCOMES:
Functional/Structural brain changes | Prior to intervention and after 6 months of intervention
Plasma biomarkers | Prior to intervention and after 6 months of intervention
Cognitive Function based on neuropsychological test-performance | Prior to intervention and after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Neurology, Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany